CLINICAL TRIAL: NCT00401661
Title: Sexuality And Management of Benign Prostatic Hyperplasia With Alfuzosin 10mg Once Daily (XATRAL 10mg OD), Open, 24-week Study.
Brief Title: Sexuality And Management of Benign Prostatic Hyperplasia With Alfuzosin
Acronym: SAMBA-Thailand
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALFUS_L_01241
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — alfuzosin

ARMS (1):
- 1 (Experimental): Alfuzosin for 24 weeks
  Interventions: Drug: Alfuzosin

INTERVENTIONS:
Drug: Alfuzosin — One tablet of 10mg once daily at the end of evening meal

SUMMARY:
Primary objective:

* End-point improvement from baseline in Male Sexual Health Questionnaire Ejaculation domain (MSHQ-EjD)in men with lower urinary tract symptoms (LUTS)suggestive of benign prostatic hyperplasia (BPH) treated for 6 months with XATRAL 10mg once daily OD.

Secondary objectives:

* MSHQ-EjD improvement by visit
* Improvement in International Prostate Symptom Score (IPSS) total score, voiding and filling subscores, nocturia and bother score at end-point and by visit
* Onset of action of XATRAL 10mg OD
* Tolerability of XATRAL 10mg OD including occurrence of acute urinary retention.

ELIGIBILITY:
Inclusion criteria:

* Patients suffering from moderate to severe LUTS suggestive of BPH
* I-PSS total score ≥ 8
* Patients sexually active

Exclusion criteria:

* Known history of hepatic or severe renal insufficiency, unstable angina pectoris, concomitant life-threatening condition
* Previous prostate surgery, minimally invasive procedure within 6 months prior to inclusion. Planned prostate biopsy, prostate surgery or minimally invasive procedure during the whole study period
* Active urinary tract infection or prostatitis, neuropathic bladder, a diagnosed prostate cancer
* Treatment with 5alpha-reductase inhibitors or phytotherapy within 6 months prior to inclusion, or alpha1-blockers within 30 days prior to inclusion
* Patients receiving any treatment for erectile dysfunction (i.e. phosphodiesterase-5 inhibitors) at inclusion
* History of postural hypotension or syncope
* Known hypersensitivity to alfuzosin

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
MSHQ Ejaculation score | End of treatment

SECONDARY OUTCOMES:
MSHQ Ejaculation score | After 4 weeks of treatment
MSHQ Ejaculation score | After 12 weeks of treatment
Acute Urinary Retention | End of treatment
Correlation between MSHQ and IPSS | End of treatment
I-PSS total score | After 1 week of treatment
I-PSS total score | After 4 weeks of treatment
I-PSS total score | After 12 weeks of treatment
I-PSS total score | End of treatment
IPSS total score decrease = 3 points | End of treatment
IPSS: filling sub-score | After 1 week of treatment
IPSS: filling sub-score | After 4 weeks of treatment
IPSS: filling sub-score | After 12 weeks of treatment
IPSS: filling sub-score | End of treatment
IPSS: nocturia symptoms sub-score | After 1 week of treatment
IPSS: nocturia symptoms sub-score | After 4 weeks of treatment
IPSS: nocturia symptoms sub-score | After 12 weeks of treatment
IPSS: nocturia symptoms sub-score | End of treatment
IPSS: voiding sub-score | After 1 week of treatment
IPSS: voiding sub-score | After 4 weeks of treatment
IPSS: voiding sub-score | After 12 weeks of treatment
IPSS: voiding sub-score | End of treatment
MSHQ ejaculation: erection sub-score | After 4 weeks of treatment
MSHQ ejaculation: erection sub-score | After 12 weeks of treatment
MSHQ ejaculation: erection sub-score | End of treatment
MSHQ ejaculation: satisfaction sub-score | After 4 weeks of treatment
MSHQ ejaculation: satisfaction sub-score | After 12 weeks of treatment
MSHQ ejaculation: satisfaction sub-score | End of treatment
Quality of Life | After 4 weeks of treatment
Quality of Life | After 12 weeks of treatment
Quality of Life | End of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Natesumroeng Taweeporn, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bangkok, Thailand